CLINICAL TRIAL: NCT03361059
Title: Falling Risks in Elderly Adults: a Prospective Cohort Study
Brief Title: Falling Risks in Elderly Adults : a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Donación Francisco Santojanni (Other)
Responsible Party: Principal Investigator, Victoria Di Giorgio, Physical Therapist, Hospital Donación Francisco Santojanni
Other Study IDs: HGADFS11052017-01
Record Dates: First submitted 2017-11-10; First posted 2017-12-04 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Fall
Keywords: risk factors; elderly patients; risk of falling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: the prevalence of falls in adults aged 65 years or older living in the community is 30%, being the second cause of accidental fatal injury and the fifth cause of death. About 20 to 30% of falls result in injuries: 10% constitute serious injuries, from which 5% are fractures. As a result, older adults decrease their mobility, are afraid of falling depressed and socially isolated, increasing the risk of later falls, death and health costs. Falls and their consequences can be prevented, so knowing and assessing the demographic, medical, self-perceived and functional characteristics constitutes an important information for health professionals. Given the high rate (29.59%) of older adults treated at the Physical Therapy outpatient consult of the "Hospital Francisco Santojanni" and the relevance of falls in this population, it is convenient to take a behavior and start by knowing their risk characteristics.

Objectives: to determine the incidence of falls of adults aged 65 years and older, seen in the Physical Therapy outpatient consult of the "Hospital Francisco Santojanni"; to describe the characteristics of these population and to identify the potential risk-of-falling factors.

Subjects and Methods: observational, prospective, longitudinal cohort study. Demographic (age and sex), medical (history of falls, visual alterations, medication and walking aids), self-perceived (fear of falling and instability perception) and functional characteristics (Test of Timed up and Go, Dynamic Index of gait and balance tests) will be evaluated in those patients of 65 years or more who initiate physical treatment in the outpatient consult of the of the "Hospital Francisco Santojanni" "Autonomous City of Buenos Aires, from March 2017 to February 2018, with a follow-up of 6 months until August 2018, to verify the development of the fall event

ELIGIBILITY:
Inclusion Criteria:

* Patients of 65 years or more treated at the Physical Therapy outpatient consult of the " Hospital Francisco Santojanni" that they walk at least inside their home and have signed informed consent

Exclusion Criteria:

* patients who walk with partial body weight load
* patients using a lower limb immobilization device

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: outpatient elderly patients of 65 years or more living in the community
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
Fall | From May 2017 to August 2018
  an event that results in a change of body position that forces a person to make contact with the ground or other support surface at a lower level, unintentionally and unexpectedly, without being the consequence of an important intrinsic event (such as loss of consciousness, sudden onset of paralysis or epileptic seizure), or unavoidable external danger (such as the collapse of a chair or violent blow). The outcome variable will be measured by a phone call.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Donación Francisco Santojanni, Ciudad Autonoma de Buenos Aire, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided